CLINICAL TRIAL: NCT00003631
Title: High-Dose Chemo-Radiotherapy for Patients With Primary Refractory and Relapsed Hodgkin's Disease
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Refractory or Relapsed Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-071; CDR0000066714 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1480
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Filgrastim; Carboplatin; Carmustine; Cyclophosphamide; Cytarabine; Etoposide; Ifosfamide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

ARMS (3):
- Arm I (Experimental): (0-1 adverse prognostic factors): Patients receive ifosfamide by 24 hour infusion on day 2. Carboplatin is administered on day 2. Etoposide IV is administered once daily on days 1-3. Patients then receive filgrastim (G-CSF) subcutaneously or IV on days 5-12. Patients receive another course of ICE chemotherapy 2-3 weeks after the first course.
  Interventions: Biological: filgrastim
- Arm II (Experimental): (2 adverse prognostic factors): Patients receive the first course of ICE as in Arm I
  Interventions: Biological: filgrastim
- Arm III (Experimental): Arm III (3 adverse prognostic factors): Patients receive cyclophosphamide IV daily for 2 days, then G-CSF beginning on day 4 until blood stem cells are collected
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: etoposide; Drug: ifosfamide; Drug: melphalan; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
  Arms: Arm III
Drug: carmustine
  Arms: Arm III
Drug: cyclophosphamide
  Arms: Arm III
Drug: cytarabine
  Arms: Arm III
Drug: etoposide
  Arms: Arm III
Drug: ifosfamide
  Arms: Arm III
Drug: melphalan
  Arms: Arm III
Procedure: bone marrow ablation with stem cell support
  Arms: Arm III
Procedure: peripheral blood stem cell transplantation
  Arms: Arm III
Radiation: radiation therapy
  Arms: Arm III

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients with refractory or relapsed Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of a high-dose chemoradiotherapy regimen in patients with refractory or relapsed Hodgkin's lymphoma.

OUTLINE: Patients are stratified into 1 of 3 treatment arms (0-1 adverse prognostic factors vs 2 adverse prognostic factors vs 3 adverse prognostic factors).

* Arm I (0-1 adverse prognostic factors): Patients receive ifosfamide by 24 hour infusion on day 2. Carboplatin is administered on day 2. Etoposide IV is administered once daily on days 1-3. Patients then receive filgrastim (G-CSF) subcutaneously or IV on days 5-12. Patients receive another course of ICE chemotherapy 2-3 weeks after the first course.

Leukapheresis is performed once WBC reaches at least 3000/mm^3 and continues until enough peripheral blood stem cells are collected.

Patients who have never received prior radiotherapy will receive accelerated hyperfractionated total lymphoid irradiation (TLI) twice a day for 5 days (days -10 to -6). Cyclophosphamide IV is then administered on days -5 and 4. Etoposide IV is administered by continuous infusion over 4 days (days -5 to -2).

Patients who have had prior radiotherapy receive high dose chemotherapy. Cyclophosphamide IV is administered on days -6 and -5. Etoposide IV is administered by continuous infusion over 4 days (days -6 to -3). Carmustine IV is administered on day -2.

Peripheral blood stem cells are infused 24-36 hours after high-dose chemotherapy. G-CSF is administered beginning on day 1 and continuing until blood counts recover.

* Arm II (2 adverse prognostic factors): Patients receive the first course of ICE as in Arm I.

Apheresis is performed once WBC is greater than 3000/mm^3 and continues until enough cells are collected. The second course of ICE is then administered.

Ifosfamide is administered by 48 hour continuous infusion on days 1-2. Carboplatin is administered on day 3. Etoposide IV is administered every 12 hours for 3 doses beginning on day 1. Patients receive G-CSF on days 5-14.

Patients who have never received prior radiotherapy will receive accelerated hyperfractionated TLI for 5 days (days -10 to -6). Cyclophosphamide IV is then administered every 12 hours on days -5 to -2. Etoposide IV is administered by continuous infusion over 4 days (days -5 to -2).

Patients who have had prior radiotherapy receive high-dose chemotherapy. Cyclophosphamide IV is administered every 12 hours on days -6 to -3. Etoposide IV is administered by continuous infusion over 4 days (days -6 to -3). Carmustine IV is administered on day -2.

Peripheral blood stem cells are infused 24-36 hours after high dose chemotherapy. G-CSF is administered beginning on day 1 and continuing until blood counts recover.

* Arm III (3 adverse prognostic factors): Patients receive cyclophosphamide IV daily for 2 days, then G-CSF beginning on day 4 until blood stem cells are collected.

Patients then undergo apheresis until enough cells are collected.

Patients receive high-dose chemotherapy. Ifosfamide IV is administered for 1 hour. Etoposide is administered by continuous infusion for 12 hours. Carboplatin IV is administered for 1 hour. Etoposide is again administered by continuous infusion for 12 hours. Treatment is repeated daily for 5 days.

Peripheral blood stem cells are reinfused 24-36 hours after the last dose of chemotherapy. G-CSF is administered beginning on day 1 and continuing until blood counts recover.

Patients who have never received prior radiation will now receive accelerated hyperfractionated TLI twice daily for 5 days. Patients receive a second course of high dose chemotherapy 45-90 days after reinfusion of cells. Etoposide IV and cytarabine IV are administered every 12 hours for 4 days (days -6 to -3). Melphalan IV is administered on day -2.

Patients who have received prior radiation therapy receive a second course of high-dose chemotherapy. Carmustine IV is administered on day -7. Etoposide IV and cytarabine IV are administered every 12 hours for 4 days (days -6 to -3). Melphalan IV is administered on day -2.

Peripheral blood stem cells are reinfused 24-48 hours after completion of second course chemotherapy. G-CSF is administered beginning on day 1 and continuing until blood counts recover.

Patients are followed every 3 months for the first 2 years, every 4 months during years 3-5, and every 6 months thereafter.

PROJECTED ACCRUAL: This study will accrue 80 patients within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed residual or relapsed Hodgkin's lymphoma following conventional dose standard chemotherapy
* Presence of the following prognostic factors are allowed:

  * B symptoms (fever, weight loss, night sweats)
  * Extranodal disease
  * Complete remission of less than 1 year duration

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL unless history of Gilbert's disease
* No chronic active or persistent hepatitis

Renal:

* No history of chronic renal insufficiency
* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months
* No unstable angina
* No significant cardiac arrhythmias other than chronic atrial fibrillation
* Ejection fraction at least 50%

Pulmonary:

* DLCO at least 50%

Other:

* No uncontrolled infection
* HIV negative
* At least 5 years since prior malignancy except:

  * Curatively treated cutaneous basal cell carcinoma
  * Carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile women must use effective contraception

PRIOR CONCURRENT THERAPY:

* Must have failed conventional dose standard chemotherapy

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 1998-08; Primary Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Yahalom, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A - Favorable Prognostic Group | Group B - Intermediate Prognostic Group | Group C - Unfavorable Prognostic Group
Started | 50 | 44 | 24
Completed | 47 | 43 | 15
Not Completed | 3 | 1 | 9
Not completed — Patient not treated | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Evaluable for toxicity only | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Favorable Prognostic Group | Group B - Intermediate Prognostic Group | Group C - Unfavorable Prognostic Group | Total
Number analyzed (Participants) | 50 | 44 | 24 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 49 | 43 | 23 | 115
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 10 | 58
  Male | 26 | 20 | 14 | 60

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Determine the overall objective response. CR rate [as measured from the start of ICE, (or high dose CTX) to the end of transplant for those who receive it, or the end of ICE for those who do not].Complete response (CR): No evidence of Hodgkin's disease determined clinically, radiologically or pathologically when indicated
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Group A - Favorable Prognostic Group | Group B - Intermediate Prognostic Group | Group C - Unfavorable Prognostic Group
Number analyzed (Participants) | 47 | 43 | 15
participants
  Failure | 3 | 6 | 3
  Minor Response (MR) | 2 | 1 | 0
  Partial Response (PR) | 1 | 2 | 4
  Progression Free (P-Free) | 41 | 31 | 7
  Complete Response (CR) | 0 | 2 | 1
  Progression of Disease (POD) | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Group A - Favorable Prognostic Group | Group B - Intermediate Prognostic Group | Group C - Unfavorable Prognostic Group
Serious Adverse Events (participants affected / at risk) | 2/50 | 6/44 | 5/24
Other Adverse Events (participants affected / at risk) | 50/50 | 44/44 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Favorable Prognostic Group (N=50) | Group B - Intermediate Prognostic Group (N=44) | Group C - Unfavorable Prognostic Group (N=24)
Cardiac ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (General disorders) | 1 (1) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Supravent arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
GI, other (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Favorable Prognostic Group (N=50) | Group B - Intermediate Prognostic Group (N=44) | Group C - Unfavorable Prognostic Group (N=24)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 10 (10) | 3 (3) | 4 (4)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 46 (46) | 41 (41) | 23 (23)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (21) | 14 (14) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 20 (20) | 12 (12) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 32 (32) | 16 (16) | 8 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 30 (30) | 25 (25) | 11 (11)
Leukocytes (Blood and lymphatic system disorders) | 46 (46) | 41 (41) | 23 (23)
Lymphopenia (Blood and lymphatic system disorders) | 49 (49) | 43 (43) | 23 (23)
Neutrophils (Blood and lymphatic system disorders) | 46 (46) | 40 (40) | 22 (22)
Platelets (Blood and lymphatic system disorders) | 46 (46) | 39 (39) | 23 (23)
Pneumonitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
SGOT (AST) (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 2 (2)
SGPT (ALT) (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes